CLINICAL TRIAL: NCT00974103
Title: Persistent Low Back Pain and Pelvic Pain 3-6 Months Post Partum
Brief Title: Persistent Low Back and Pelvic Pain 3-6 Months Post Partum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University of Stavanger (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/798; 2009/798 (Other: Regional Ethics Committee)
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Pelvic Girdle Pain Post Partum; Low Back Pain Post Partum
Keywords: low back pain; pelvic pain; pelvic girdle pain; post partum
MeSH Terms: conditions — Low Back Pain; Pelvic Pain; Pelvic Girdle Pain | interventions — Pregnancy; Exercise; Postpartum Period; Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chiropractic treatment, exercise (Experimental): Chiropractic treatment and exercise
  Interventions: Other: chiropractic treatment and exercises
- Exercises (Experimental): Exercise advise
  Interventions: Other: exercise advise

INTERVENTIONS:
Other: exercise advise — Exercises
  Other Names: Pregnancy; Back pain; Exercise; Post partum; chiropractic
  Arms: Exercises
Other: chiropractic treatment and exercises — Manipulation, mobilisation, soft tissue work, ergonomic and exercise advise. Maximum 12 treatments
  Other Names: Manipulation; Pregnancy; Back pain; Exercise; Post partum; chiropractic
  Arms: Chiropractic treatment, exercise

SUMMARY:
The purpose of this study is to identify how many females have persistent low back pain and/or pelvic pain 3-6 months post partum. The females that have persistent pelvic pain can continue in the study and be examined by a chiropractor. They will then divide the females into Hanne Alberts 5 subgroups of pelvic pain. The females that have one-sided pelvic pain will be invited to participate in a randomised controlled study where chiropractic intervention is compared to exercises.

DETAILED DESCRIPTION:
The study is a follow up study to "Prevalence of low back pain and pelvic pain in the pregnant population in Stavanger".

ELIGIBILITY:
Inclusion Criteria:

* Low back and\or pelvic girdle pain during pregnancy
* Fluent understanding of spoken and written Norwegian

Exclusion Criteria:

* hospitalisation due to pain or complications post partum

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 20 weeks after the initial assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jan P Larsen, MD Dr med, Study Director — Helse Stavanger HF
Locations (1):
- Stavanger university hospital, Stavanger, Norway